CLINICAL TRIAL: NCT02976623
Title: Effects of Metric-based Feedback Training on Acquisition of Sonographic Skills Relevant to Performance of Ultrasound Guided Axillary Brachial Plexus Block
Brief Title: Metric-based Feedback Training for the Acquisition of Sonographic Skills
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College Cork (Other)
Responsible Party: Principal Investigator, Brian Declan O'Donnell, Consultant Anaesthetist, Senior Lecturer, University College Cork
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: ECM 4 (f) 19/01/16
Record Dates: First submitted 2016-11-11; First posted 2016-11-29 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Simulation Training
Keywords: metrics; feedback; ultrasound-guided; procedural skills

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- feedback group (Other): this group will receive the intervention "metric-based feedback training" on their performance. this will be based on validated metrics and errors, a trained investigator will deliver this feedback. It will be accompanied by deliberate practice
  Interventions: Other: metric-based feedback training
- control group (No Intervention): this control group will receive a standard type feedback on their performance "no intervention". It will be delivered by a consultant anaesthetist who will be instructed to deliver feedback as they ordinarily do during their clinical practice

INTERVENTIONS:
Other: metric-based feedback training — Structured feedback; a trained investigator will give feedback according to a set of metrics and errors previously developed and validated. Trainees will undergo deliberate practice on the volunteer until they demonstrate adequate and objective performance as assessed by the set of metrics and errors provided.
  Arms: feedback group

SUMMARY:
The investigators hypothesized that feedback based on previously developed and validated metrics will improve novices' learning of procedural skills.

The objective of this study was to determine the effect of a structured, objective and terminal feedback on novices' performance skills of ultrasonography part of ultrasound-guided axillary brachial plexus block.

DETAILED DESCRIPTION:
The use of ultrasound guidance during performance of peripheral nerve blocks improves success rate, shortens performance time and reduces the risk of inadvertent vascular puncture. Safe and effective procedure performance requires the operator to make a series of real-time, high stakes decisions relevant to interpretation of sonographic anatomy and subsequent nerve visualization, needle-to-nerve guidance, needle-to-nerves approximation and local anesthetic deposition. Teaching novices to perform ultrasound-guided nerve blocks should include rendering and assessment of its component skills such as interpretation of sonographic anatomy, consistent needle imaging and correct placement of local anesthetics. Learning and teaching ultrasound-related motor skills is challenging within the current landscape of medical and training education. Simulated learning has been advocated as it can facilitate deliberate practice as opposed to repeated practice. Simulation and e-learning are flexible training modalities, which facilitate procedural skills rehearsal in a safe environment, free from risk to patients, and permitting real time feedback. Deliberate practice with feedback in a simulated environment may accelerate the rate of skill acquisition. Feedback is a predictor of effective learning and a useful tool for novices learning new skill. However summative feedback is superior to concurrent feedback for procedural skill acquisition during simulated but not clinical training and for skill retention. The characteristics of feedback, which influence its effect on learning, include timing, content, who initiates (elicits) it and the format and motivation applied to its delivery. Feedback positively influences skill acquisition by novice learners. How trainees adopt objective versus subjective feedback remained largely undetermined. The investigators hypothesize that feedback based on previously developed and validated metrics will improve novices' learning of procedural skills.

The objective of this study was to determine the effect of a structured, objective and terminal feedback on novices' performance skills of ultrasonography part of ultrasound-guided axillary brachial plexus block.

Methods:

With institutional ethical approval and having obtained written informed consent from each, 12 anesthesia trainees will be invited to participate in this prospective, randomized and blinded study.

Inclusion criteria:

i. trainees in the Irish national anesthesia training program allocated to Cork teaching hospital (CUH) ii. have performed no more than 5 ultrasound-guided peripheral nerve blocks at the time of participation.

Each participant will answer tests to ascertain visuospatial and perceptual abilities (card rotation, cube comparisons and map planning tests).

Each participant will provide baseline information prior to participation i) age ii) gender iii) handedness iv) Years since graduating from medical school v) number or estimated number of previously performed ultrasound-guided interventional procedures including securing vascular access vi) courses/workshops in ultrasound-guided procedural interventions.

All participants will receive a standard learning in the form of i) a one hour didactic lecture delivered by a single investigator which outlines basic sonographic anatomy, ultrasound physics and anatomy relevant to performing ultrasound-guided axillary brachial plexus block.

Within 24 hours of completing the learning phase, participants will be asked to perform ultrasonography of left axilla of a volunteer. This will be followed by either feedback A or feedback B (based on random allocation). Feedback will terminal, summative and commence five minutes after each participant completed the tasks.

Task description:

1. Participant perform ultrasonography of left axilla and adjacent upper limb as if preparing to perform ultrasound-guided axillary brachial plexus block
2. Participant identify the four terminal branches of the brachial plexus; identify each on the screen by using the pointer provided (or freeze image and use arrow on the screen) and name each verbally.
3. Participant identify the adjacent structures/vessels relevant to the block by indicating them individually using the pointer provided (or freeze image and use arrow on the screen) and name each verbally.
4. Once participant have obtained an optimal ultrasound image, participant is requested to indicate the intended needle insertion point on the skin using the pointer provided.

Participants will be provided with an opportunity to practice performing the tasks for up to 30 minutes. Within one hour of completing the feedback session, participants will be asked to attempt the same tasks again. Performance before and after feedback delivered will be video-recorded according to a predefined protocol by a trained investigator. Imaging will be obtained by an investigator using a handheld camera. Concurrent ultrasound video images will be recorded using the Digital Video Recorder (DVR) feature of the Ultrasonics Tablet (Sonix Design Centre, B.K Ultrasound, Richmond, Canada). All video recordings will be edited using a video editing software (Apple Movie, version 10.0.5, Apple Computer Inc. USA) to present the procedure together with the ultrasound output on one screen

Types of Feedback:

i. Feedback A: Standard feedback; a consultant anesthetists will be asked to give feedback as would normally give during performance of such a task in a clinical situation.

ii. Feedback B: Structured feedback; a trained investigator will give feedback according to a set of metrics and errors previously developed and validated. Trainees will undergo deliberate practice on the volunteer until they demonstrate adequate and objective performance as assessed by the set of metrics and errors provided.

Video assessment and scoring:

Two trained, independent and blinded assessors will score the video recordings for a set of metrics and errors previously developed and validated. The number of steps completed and errors committed will be compared for i) Group defined by preceding type of feedback, ii) Pre versus post for each feedback session

ELIGIBILITY:
Inclusion Criteria:

* Anaesthesia trainees in the first two years of training at Cork University Hospital
* having performed no more than 5 ultrasound-guided peripheral nerve blocks

Exclusion Criteria:

* refusal to consent
* have performed more than 5 ultrasound-guided peripheral nerve blocks

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2016-06; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
number of steps completed and number of errors committed | through study completion, an average of one year

SECONDARY OUTCOMES:
scanning time | through study completion, an average of one year
  time elapsed from placement of ultrasound probe on volunteer to the time of identification of needle insertion point

CONTACTS AND LOCATIONS:
Locations (1):
- Cork University Hospital, Cork, Ireland

IPD SHARING:
Plan to Share IPD: No